CLINICAL TRIAL: NCT00040560
Title: Study of 111In-DAC as an Medical Imaging Agent for Lung Cancer and Brain Cancer Consistent With Metastatic Lung Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Copharos (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CP102
Record Dates: First submitted 2002-06-28; First posted 2002-07-02 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-01

CONDITIONS: Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Brain Neoplasms; Metastases, Neoplasm
Keywords: Lung Cancer; Metastatic Brain Cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Brain Neoplasms; Neoplasm Metastasis

INTERVENTIONS:
Drug: 111In-DAC
Procedure: Diagnostic

SUMMARY:
The purpose of this study is to investigate the safety and imaging ability of 111In-DAC when used with planar and SPECT imaging for the detection of lung cancer and brain cancer consistent with metastatic lung cancer.

ELIGIBILITY:
Inclusion Criteria

Patients will be eligible for the study if they:

* Are male or non-pregnant, non-lactating females 18 years of age or older (must agree to use an appropriate and effective method of birth control during the study and for 2 weeks after study)
* Have an ECOG performance status of Zero or One
* Are being evaluated for known or suspected non-small-cell lung cancer (NSCLC), or known brain lesions consistent with metastatic lung cancer
* (For NSCLC patients)Have been previously scheduled for biopsy or surgical excision of the suspected NSCLC, or have a pathological diagnosis of lung cancer within 2 months of enrollment but have received no previous treatment
* (For brain cancer patients) Have clinical signs and symptoms consistent with a primary NSCLC with histological or cytopathological confirmation. Patients cannot have received previous treatment with radiation to the brain.
* Have signed an informed consent form

Exclusion Criteria

Patients will not be eligible for this study if they:

* Have a history or suspicion of significant allergic reaction or anaphylaxis to any of the 111In-DAC components
* Have a clinically unstable medical condition or opportunistic infection, a life-threatening disease state, impaired renal or hepatic function or are immunosuppressed
* Are taking or have taken part in any investigational study within 30 days of start of study
* Have received an indium agent within 30 days of start of study
* Are not able to remain immobile during scanning time
* Have taken drugs that may damage the kidneys within 2 weeks of start of study
* Have abnormal laboratory test results: hemoglobin<9.5 gms/dl, serum creatinine>1.5mg/100ml, alkaline phosphatase 2X the upper limit of normal
* Have undergone an excisional and/or needle localization biopsy within 4 days prior to study drug administration
* Have undergone a PET scan within 7 days prior to study drug administration
* Have any active or previously treated second malignancy except carcinoma in situ of the uterine cervix or non-melanoma skin cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Sutter Roseville Medical Center, Roseville, California
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida